CLINICAL TRIAL: NCT01180634
Title: A Phase 3, Multi-Center, Multinational, Randomized, Double-Blind, Placebo-Controlled Study To Evaluate The Efficacy And Safety Of MP-376 (Levofloxacin Inhalation Solution; Aeroquin™) In Stable Cystic Fibrosis Patients
Brief Title: MP-376 (Aeroquin™, Levofloxacin for Inhalation) in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mpex-207; 2010-019515-38 (EudraCT Number)
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Results first posted 2024-04-30 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aeroquin 240 mg (Experimental): Participants received 240 milligrams (mg) of Aeroquin by inhalation route twice daily (BID) for a period of 28 days.
  Interventions: Drug: Aeroquin
- Placebo (Placebo Comparator): Participants placebo matching Aeroquin by inhalation route, BID for a period of 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aeroquin — Inhalation Solution
  Other Names: MP-376, Levofloxacin Inhalation solution 240 mg
  Arms: Aeroquin 240 mg
Drug: Placebo — Inhalation Solution
  Arms: Placebo

SUMMARY:
Patients with cystic fibrosis (CF) suffer from chronic infections of the lower respiratory tract that can be caused by one or multiple bacteria, including Pseudomonas aeruginosa, which has been particularly problematic to eradicate and been implicated as the major cause of morbidity and mortality in CF patients. Aerosol delivery of antibiotics directly to the lung increases the local concentrations of antibiotic at the site of infection resulting in improved antimicrobial effects compared to systemic administration. Decreased efficacy, intolerance and high treatment burden with currently available therapies indicate a need for additional therapies. MP-376 (Aeroquin™) is a novel formulation of the fluoroquinolone levofloxacin that has been optimized for aerosol delivery. Preclinical and clinical studies conducted to date show that aerosol doses of MP-376 are safe and well tolerated, exert an antimicrobial effect, improve lung function and reduce the need for other anti-pseudomonal antibiotics. High concentrations of levofloxacin in the lung delivered as MP-376 are active against CF pathogens including those with high minimum inhibitory concentration (MIC) levels to aminoglycosides such as tobramycin (TOBI®) and other inhaled antimicrobial agents. Inhaled MP-376 can be delivered rapidly and efficiently using a customized PARI investigational configuration of the eFlow® nebulizer system.

DETAILED DESCRIPTION:
This trial will be a double-blind, placebo-controlled study to evaluate the efficacy and safety of levofloxacin administered as MP-376 given for 28 days by the aerosol route to CF patients.

Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria (selected):

* >/= 12 years of age
* Confirmed Diagnosis of Cystic Fibrosis
* Positive sputum culture for P. aeruginosa at screening and within the past 12 months
* Patients are able to elicit an FEV1 >/= 25% but </= 85% of predicted value at screening
* Have received at least 3 courses of inhaled antimicrobials over the preceding 12 months
* Clinically stable with no changes in health status within the last 28 days
* Able to reproducibly produce sputum and perform spirometry

Exclusion Criteria (selected):

* Use of any nebulized or systemic antibiotics within 28 days prior to baseline
* History of hypersensitivity to fluoroquinolones or intolerance with aerosol medication
* Evidence of respiratory infections within 14 days prior to dosing
* CrCl < 20ml/min or < 20ml/min/1.73 m2 at Screening

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2010-11-04 (Actual); Primary Completion 2012-05-07 (Actual); Study Completion 2012-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (103):
- United States (86):
  - Mobile, Alabama
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Tucson, Arizona
  - La Jolla, California
  - Long Beach, California
  - Childrens Hospital, Los Angeles, California
  - Los Angeles, California
  - Oakland, California
  - Orange, California
  - Palo Alto, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Denver, Colorado
  - Hartford, Connecticut
  - Wilmington, Delaware
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Glenview, Illinois
  - Niles, Illinois
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Portland, Maine
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Minneapolis, Minnesota
  - Jackson, Mississippi
  - Columbia, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Manchester, New Hampshire
  - Livingston, New Jersey
  - Long Branch, New Jersey
  - Morristown, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - New York, New York
  - Syracuse, New York
  - Valhalla, New York
  - Chapel Hill, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Sioux Falls, South Dakota
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Colchester, Vermont
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Portsmouth, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Australia (9):
  - John Hunter Hospital, New South Wales, New South Wales
  - Westmead Chilren's Hospital, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Mater Miscericordiae Hospital, Brisbane, Queensland
  - Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Children's Hospital, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Monash Medical Center, Melbourne
- Canada (3):
  - Hamilton, Ontario
  - Kingston, Ontario
  - Ottawa, Ontario
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center Mount Scopus, Jerusalem
  - Schneider Childrens Medical Center of Israel, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Auckland Hospital, Auckland, New Zealand

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aeroquin 240 mg | Placebo
Started | 220 | 110
Completed | 210 | 109
Not Completed | 10 | 1
Not completed — Adverse Event | 4 | 1
Not completed — Miscellaneous | 2 | 0
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Aeroquin 240 mg: Participants received 240 mg of Aeroquin by inhalation route, BID for a period of 28 days.
- Total: Total of all reporting groups
Arm/Group | Aeroquin 240 mg | Placebo | Total
Number analyzed (Participants) | 219 | 110 | 329
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (10.34) | 28.8 (10.94) | 29.2 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 47 | 152
  Male | 114 | 63 | 177
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 19
  Not Hispanic or Latino | 209 | 101 | 310
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 212 | 100 | 312
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to an Exacerbation
Description: The start of the exacerbation was determined by the earliest date at which a participant concurrently met at least 4 of the 12 modified Fuchs symptoms/signs; discontinued from the study early; died; or received an antipseudomonal agent for an event that did not meet modified Fuchs criteria but was determined to be an exacerbation by the Blinded Exacerbation.
  Fuchs symptoms/signs;
  * Change in sputum
  * New or increased hemoptysis
  * Increased cough
  * Increased dyspnea
  * Malaise, fatigue or lethargy
  * Temperature above 38oC
  * Anorexia or weight loss
  * Sinus pain or tenderness
  * Change in sinus discharge
  * Change in physical examination of the chest
  * Decrease in pulmonary function by 10 percent or more from a previously recorded value
  * Radiographic changes indicative of pulmonary infection
  Median and 95%Ci were estimated using Kaplan Meier estimates.
Time Frame: Baseline to end of study (up to 59 days)
Population: Intent-to-treat (IIT) population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Aeroquin 240 mg | Placebo
Number analyzed (Participants) | 220 | 110
Days | 58 [52 to NA] — Upper bound of 95% CI was not estimable due to low number of events | 51.5 [43 to NA] — Upper bound of 95% CI was not estimable due to low number of events
Statistical Analysis 1: Comparison: Aeroquin 240 mg vs Placebo; Test type: Superiority; p = 0.0715, Log Rank — P-value is determined using a log-rank test stratified by region (US, non-US), age (12-18 years, >18 years), and baseline FEV1 (<55%, >=55%); Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.96 to 1.84] — Hazard ratio is obtained from a Cox proportional hazards regression model adjusting for region (US, non-US), age (12-18 years, >18 years), and baseline FEV1 (<55%, >=55%)

2. Secondary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in One Second (FEV1)
Description: FEV1 was the volume of air exhaled in first second of a forced expiration as measured by spirometer. Least squares (LS) mean and standard error are determined from a repeated measures model with terms for treatment, visit, treatment*visit, region (US, non-US), age (12-18 years, >18 years), and baseline FEV1 (<55%, >=55%).
Time Frame: Baseline, day 28
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percent Predicted FEV1
Arm/Group | Aeroquin 240 mg | Placebo
Number analyzed (Participants) | 220 | 110
Percent Predicted FEV1 | 0.08 (0.638) | 1.49 (0.531)
Statistical Analysis 1: Comparison: Aeroquin 240 mg vs Placebo; Test type: Superiority; p = 0.0213, Repeared Measures Model; LSMean difference = 1.41, 95% CI 2-sided [0.21 to 2.60] — Estimates are determined from a repeated measures model with terms for treatment, visit, treatment*visit, region (US, non-US), age (12-18 years, >18 years), and baseline FEV1 (<55%, >=55%)

3. Secondary Outcome: Change From Baseline in Pseudomonas Aeruginosa Sputum Density
Description: Pseudomonas aeruginosa density was measured as log10 colony-forming units [CFU] per gram sputum. LSMean and standard are determined from a repeated measures model with terms for treatment, visit, treatment*visit, region (US, non-US), age (12-18 years, >18 years), baseline FEV1 (<55%, >=55%), and baseline organism log density.
Time Frame: Baseline, Day 28
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: log10 CFU/g
Arm/Group | Aeroquin 240 mg | Placebo
Number analyzed (Participants) | 220 | 110
log10 CFU/g | 0.04 (0.170) | -0.59 (0.139)
Statistical Analysis 1: Comparison: Aeroquin 240 mg vs Placebo; Test type: Superiority; p = 0.0002, Repeated Measures Model; LSMean difference = -0.63, 95% CI 2-sided [-0.95 to -0.30] — Estimates are determined from a repeated measures model with terms for treatment, visit, treatment*visit, region (US, non-US), age (12-18 years, >18 years), baseline FEV1 (<55%, >=55%), and baseline organism log density

4. Secondary Outcome: Change From Baseline in the Respiratory Domain of the Cystic Fibrosis Questionnaire Revised (CFQ-R)
Description: The Cystic Fibrosis Questionnaire (CFQ-R) is a disease-specific instrument that measures health-related quality of life (HRQOL) for adolescents and adults with cystic fibrosis (CF). Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. LSMean and standard error were determined from a repeated measures model with terms for treatment, visit, treatment*visit, region (US, non-US), age (12 to 18 years, > 18 years), Baseline FEV1 (<55%, ≥ 55%), and Baseline value.
Time Frame: Baseline, Day 28
Population: ITT population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Aeroquin 240 mg | Placebo
Number analyzed (Participants) | 218 | 108
Score on a scale | 4.66 (1.374) | 4.94 (1.118)
Statistical Analysis 1: Comparison: Aeroquin 240 mg vs Placebo; Test type: Superiority; p = 0.8335, Repeated Measures Model; LSMean difference = 0.28, 95% CI 2-sided [-2.30 to 2.85] — Estimates were determined from a repeated measures model with terms for treatment, visit, treatment*visit, region (US, non-US), age (12 to 18 years, > 18 years), Baseline FEV1 (<55%, ≥ 55%), and Baseline value

5. Secondary Outcome: Relative Change From Baseline in Percent Predicted FEV1
Description: as for outcome 2
Time Frame: Baseline, Day 28
Population: ITT population with available data at specific timepoint.
Measure: Least Squares Mean (Standard Error); unit: Percent Predicted FEV1
Arm/Group | Aeroquin 240 mg | Placebo
Number analyzed (Participants) | 218 | 109
Percent Predicted FEV1 | 1.24 (1.041) | 3.66 (0.866)
Statistical Analysis 1: Comparison: Aeroquin 240 mg vs Placebo; Test type: Superiority; p = 0.0122, Repeated Measures Model; LSMean difference = 2.42, 95% CI 2-sided [0.53 to 4.31]

6. Secondary Outcome: Time to Administration of Other Systemic and/or Inhaled Antipseudomonal Antimicrobials
Description: Participants who had at least one of four worsening respiratory symptoms (increased cough, increased sputum/chest congestion, decreased exercise tolerance, decreased appetite) at the time of administration of the anti-pseudomonal antimicrobial agent were included in the analysis. Median and 95% CI are estimated using Kaplan Meier estimates.
Time Frame: Baseline to end of study (up to 59 days)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Aeroquin 240 mg | Placebo
Number analyzed (Participants) | 220 | 110
Days | 59 [53 to 60] | 55 [43 to NA] — Upper bound of 95% CI was not estimable due to low number of events
Statistical Analysis 1: Comparison: Aeroquin 240 mg vs Placebo; Test type: Superiority; p = 0.3000, Log Rank — [p-value comment as in outcome 1, analysis 1]; Cox Proportional Hazard = 0.82, 95% CI 2-sided [0.60 to 1.12] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Time to First Hospitalization
Description: Median and 95%CI was estimated using Kaplan Meier estimates.
Time Frame: Baseline to end of study (up to 59 days)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Aeroquin 240 mg | Placebo
Number analyzed (Participants) | 220 | 110
Days | NA [60 to NA] — Median and upper bound of confidence interval were not estimable due to low number of events. | NA [NA to NA] — Median, lower and upper bound of confidence interval were not estimable due to low number of events.
Statistical Analysis 1: Comparison: Aeroquin 240 mg vs Placebo; Test type: Superiority; p = 0.8670, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.47 to 2.04] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An AE was defined as any unfavorable or unintended sign, symptom, or disease temporally associated with the use of a Study Drug, whether or not considered related to the Study Drug.
  An AE could potentially be a new disease, any untoward event, or an exacerbation of a pre-existing condition. AEs included, but were not limited to:
  * Any symptom not previously reported by the patient (medical history)
  * An exacerbation of a pre-existing illness
  * An increase in frequency or intensity of a pre-existing episodic event or condition
  * A condition first detected or diagnosed after Study Drug administration even though the condition may have been present before the start of the study
  * Overdose of Study Drug
Time Frame: From start of study until end of study (Up to 59 days)
Population: Safety population included all randomized participants in the study who received at least 1 dose of study drug or placebo.
Measure: Number; unit: participants
Arm/Group | Aeroquin 240 mg | Placebo
Number analyzed (Participants) | 219 | 110
participants | 214 | 108

ADVERSE EVENTS:
Time Frame: From start of study until end of study (Up to 59 days)
Description: Safety Population
Arm/Group | Aeroquin 240 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/219 | 0/110
Serious Adverse Events (participants affected / at risk) | 21/219 | 11/110
Other Adverse Events (participants affected / at risk) | 207/219 | 106/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aeroquin 240 mg (N=219) | Placebo (N=110)
Disease progression (General disorders) | 15 (15) | 11 (11)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aeroquin 240 mg (N=219) | Placebo (N=110)
Nausea (Gastrointestinal disorders) | 14 | 1
Nausea (General disorders) | 92 | 42
Exercise tolerance decreased (General disorders) | 28 | 11
Exercise tolerance decreased (General disorders) | 42 | 22
Pyrexia (General disorders) | 16 | 2
Pyrexia (Infections and infestations) | 10 | 6
Forced expiratory volume decreased (Investigations) | 21 | 10
Weight decreased (Investigations) | 36 | 21
Decreased appetite (Metabolism and nutrition disorders) | 22 | 12
Dysgeusia (Nervous system disorders) | 77 | 0
Headache (Nervous system disorders) | 14 | 3
Sinus Headache (Nervous system disorders) | 26 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 124 | 51
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 26 | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 35 | 10
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 44 | 21
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 37 | 18
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 12 | 4
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 67 | 39
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 23 | 15
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 91 | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other